CLINICAL TRIAL: NCT07173764
Title: Congenital and Maternal Point of Care Rapid Testing for Syphilis Study, Uganda
Acronym: COMPARTS
Status: Not yet recruiting | Type: Observational
Sponsor: St George's, University of London (Other)
Collaborators: Johns Hopkins University (Other); MU-JHU CARE (Other)
Responsible Party: Sponsor
Other Study IDs: 2025.0124
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Syphilis; Syphilis, Congenital
Keywords: syphilis; point of care test
MeSH Terms: conditions — Syphilis; Syphilis, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
Syphilis is an infection which affects about 1 in 25 pregnant women in Uganda. If the infection is not diagnosed and treated this can be a risk to the mother and unborn baby's health. This study aims to see whether a new test for syphilis infection in mothers and babies which can give a result in 10 minutes is as good as the standard tests that are done in the laboratory and take hours or days to provide results.

DETAILED DESCRIPTION:
Maternal syphilis is a major cause of poor birth outcomes including congenital syphilis (CS), which may cause miscarriage, stillbirth, or birth defects. In 2016, the global maternal syphilis prevalence was an estimated 0.69% resulting in a global CS rate of 473 per 100,000 live births and 661,000 total CS cases, including 355,000 adverse birth outcomes and 306,000 non-clinical CS cases (infants without clinical signs born to untreated mothers). The prevalence of syphilis and CS in Uganda is high. In a study of 570 antenatal women with HIV in Kampala, 5.1% had syphilis. Other Ugandan studies have demonstrated >3% prevalence of antenatal syphilis and CS prevalence of 3.8% among newborns.

Testing for syphilis in pregnancy accompanied by effective treatment with benzyl penicillin G (benzathine penicillin) can significantly reduce the risk of CS. This should ideally occur as early in pregnancy as possible, with each additional week of delay in diagnosis and treatment increasing the risk of CS. Syphilis testing in Uganda, as in many other low- and middle-income countries, primarily relies on rapid diagnostic tests that detect IgG antibodies against Treponema pallidum, the bacterium responsible for syphilis. These treponemal tests (TT) are highly sensitive and therefore valuable for initial diagnosis but cannot differentiate between untreated and previously treated syphilis due to their lifelong positive result.

To confirm infection, a lipoidal, non-treponemal test (NTT) like the rapid plasma reagin (RPR) test is also required. NTTs are relatively inexpensive but require a reliable electricity supply, reagents, laboratory infrastructure and trained laboratory personnel. The performance of tests like the RPR may be suboptimal with wide inter-laboratory variation, especially in low-income settings with high humidity levels. This prevents diagnosis and treatment from occurring during the same antenatal visit, leading to treatment delays or treatment being missed entirely. Following treatment, NTT antibody titres are ideally followed up to 12 or 24 months (depending on syphilis stage and HIV status), which is also complicated by the above issues.

In babies born to mothers with syphilis, serological diagnosis of CS is made by demonstrating a ≥4- fold higher NTT titre in infant compared to maternal blood (e.g., maternal NTT titre 1:2, infant NTT titre 1:8). The higher titre in the infant suggests that NTT antibodies were being made in the fetus representing infant infection. TTs are not useful in the serological diagnosis of CS because they likely represent transplacental transfer of maternal treponemal IgG. The infrastructure required and delays to provision of results for traditional RPR testing creates similar challenges in diagnosing and treating infants born at risk of CS or with clinical features consistent with CS as it does in pregnant persons.

Lateral flow assays are simple, quick, and potentially low-cost tests that can be conducted at the point- of-care, enabling clinicians to make timely diagnoses and allowing testing and treatment to be provided during the same encounter. This has clear benefits for patients in reducing number of clinic visits required, and in the context of the Ugandan healthcare system where only 37% of women receive antenatal care in the first trimester and 68% have 4 or more antenatal visits, reducing any delays to treatment and risk of loss to follow up are essential.

The Chembio DPP Syphilis TnT (Chembio Diagnostics, Medford, NY, USA) is a point of care test (POCT) that gives both treponemal IgG and IgM and non-treponemal IgG and IgM results. It is the second generation of a device with improvements in sensitivity of non-treponemal tests compared to the first generation Syphilis Screen & Confirm test. The results provided by the Chembio DPP TnT and the CS test (under development) could allow healthcare providers to accurately diagnose pregnant women and newborns with syphilis and commence treatment during the same clinical encounter, reducing delayed and missed treatment. It has the potential to allow for differentiation between current and past infection and is capable of quantification of treponemal and non-treponemal IgM and IgG (TnT test), and treponemal and non-treponemal IgA and IgM (CS test) which may allow improvements in the diagnosis of active infection and confirmation of treatment success.

This study will validate Chembio DPP TnT against conventional treponemal and non-treponemal testing pathways in a Ugandan population, using blood samples from pregnant women, umbilical cords, and newborns taken around the time of delivery. Validation of the Chembio DPP TnT could facilitate its implementation in streamlined diagnosis and treatment monitoring pathways that might reduce delays to treatment, improve treatment rates and confirmation of treatment success. This pilot study will demonstrate the feasibility of performing such validation in this setting and will therefore lay the groundwork for further larger studies to contribute further to this validation work.

ELIGIBILITY:
Inclusion Criteria:

* Mothers delivering at Kawempe National Referral Hospital with a positive syphilis rapid diagnostic test during their current pregnancy.

Exclusion Criteria:

* Mothers who are unable to give written informed consent.
* Mothers with evidence of neurological symptoms compatible with neurological syphilis.
* Mothers who are aged less than 14 years. Emancipated and mature minors are allowed to consent for research per Ugandan law.11
* Mothers, who in the view of the study team, are unable to adhere to required study procedures

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mothers delivering at Kawempe National Referral Hospital with a positive syphilis rapid diagnostic test during their current pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary outcomes | At enrolment
  Correlation of binary non-treponemal IgM and IgG results for the Chembio DPP Syphilis TnT with RPR positivity.
  Correlation of binary treponemal IgM and IgG results for the Chembio DPP Syphilis TnT with Treponemal Antibody (TPAB) positivity.
  Correlation of binary IgA and IgM results for the Chembio DPP Syphilis CS and Chembio DPP Syphilis TnT to the RPR results in mother and baby to confirm the diagnosis of congenital syphilis in the neonate.

CONTACTS AND LOCATIONS:
Locations (1):
- Kawempe National Referral Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No